CLINICAL TRIAL: NCT00776308
Title: Molecular Breast Imaging in the Preoperative Evaluation of Women With Biopsy Proven Breast Cancer
Brief Title: Use of Molecular Breast Imaging (MBI) to Detect Additional Disease in Women With Breast Cancer Who Are About to go to Surgery
Acronym: MBI
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Gamma Medica-Ideas (Industry)
Responsible Party: Judy Boughey, M.D., Mayo Clinic
Other Study IDs: 07-004241; NIH Grant: CA128407-01
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: molecular breast imaging; breast cancer; mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Conventional mammography is not a reliable method for determining the extent of disease in women with breast cancer. Molecular Breast Imaging (MBI) is a new nuclear medicine technique that allows the breast to be imaged in a manner similar to mammography, but without the pain of compression. Initial results with this method have shown it is very good at detecting small breast cancers (~1/4 inch).

The purpose of this study is to see if MBI is a better method than mammography in determining how much cancer is present before a woman goes to surgery.

The study will comprise 120 women with breast cancer who are going to surgery. The investigators hope that this study will demonstrate that MBI will be more accurate in determining how much cancer is present.

DETAILED DESCRIPTION:
The sensitivity of conventional mammography for evaluation of extent of disease, detection of multifocal breast cancers and contralateral breast cancers is poor. Molecular Breast Imaging (MBI) is a new nuclear medicine technique that permits the breast to be imaged in a manner similar to mammography, utilizing a Cadmium-Zinc-Telluride (CZT) gamma camera. We have developed the first dual-head MBI system in the world and preliminary results from this system indicate a high sensitivity (~90%) for the detection of breast cancers < 10mm.

The AIM of this study is to determine the sensitivity of MBI relative to mammography in the preoperative evaluation of the extent of disease in the ipsilateral and contralateral breasts in women with biopsy-proven breast cancer. We will test the HYPOTHESIS that MBI is more sensitive than mammography for preoperative evaluation and surgical planning.

The study will comprise 120 women with biopsy-proven breast cancer prior to surgery. All patients will have a diagnostic mammogram and an MBI study prior to operation. At the time of operation the pathologic findings will be correlated with both the mammogram and the MBI results.

This study will demonstrate the use of MBI in three aspects of breast cancer diagnosis: 1) detection of multifocal / multicentric disease elsewhere in the ipsilateral breast, 2) detection of contralateral breast cancer, and 3) correlation of index tumor size on MBI with pathologic size. These results may justify a role for MBI in the routine pre-operative evaluation of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Women with biopsy-proven breast cancer (invasive breast cancer or ductal carcinoma in situ)

Exclusion Criteria:

* Unable to understand and sign the consent form
* Pregnant or lactating
* Physically unable to sit upright and still for 40 minutes
* Currently receiving neoadjuvant chemotherapy or hormonal therapy
* Currently taking tamoxifen, evista (raloxifene), or an aromatase inhibitor
* Previous mastectomy
* Previous excisional biopsy of the index breast cancer

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment will be from the pool of patients undergoing surgical evaluation for breast cancer at Mayo Clinic Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2008-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The gold standard for assessing MBI will be tissue pathology. Using pathology as the gold standard, we will compare the sensitivity of MBI to that of mammography in the evaluation of this patient population. | At surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael K O'Connor, Ph.D., Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic News — http://newsblog.mayoclinic.org/2008/09/03/breast-cancer-molecular-breast-imaging-mammography/
- See also: Mayo Clinic You Tube Channel — http://www.youtube.com/watch?v=DOQBLe8MdH0